CLINICAL TRIAL: NCT05326750
Title: Non-invasive Neurostimulation as a Tool for Diagnostics and Management for Neurodegenerative Diseases
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Responsible Party: Principal Investigator, Eino Solje, MD PhD adj. prof., Kuopio University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KUH5772859
Record Dates: First submitted 2022-03-23; First posted 2022-04-14 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Alzheimer Disease; Frontotemporal Dementia; Dementia With Lewy Bodies
MeSH Terms: conditions — Alzheimer Disease; Frontotemporal Dementia; Lewy Body Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real tACS (Experimental): Four sessions (once a day, during four consecutive days) of gamma tACS (40 Hz) at 3 mA over the superior parietal cortex (Precuneus)
  Interventions: Device: Gamma tACS (40 Hz) over the superior parietal cortex
- Sham tACS (Placebo Comparator): Four sessions of sham tACS (once a day, during four consecutive days) over the superior parietal cortex (Precuneus)
  Interventions: Device: Gamma tACS (40 Hz) over the superior parietal cortex

INTERVENTIONS:
Device: Gamma tACS (40 Hz) over the superior parietal cortex — Single session of gamma tACS (40 Hz) over the superior parietal cortex

SUMMARY:
Double blinded, sham-controlled, randomized trial on repeated transcranial alternating current brain stimulation (tACS) in neurodegenerative diseases. The investigators will evaluate whether a 4-times daily repeated stimulation with gamma tACS on the posterior parietal cortex can improve symptoms in patients with neurodegenerative diseases, including dementia with Lewy Bodies, Alzheimer's disease, idiopathic normal pressure hydrocephalus and Frontotemporal dementia.

DETAILED DESCRIPTION:
Double blinded, sham-controlled, randomized trial on repeated transcranial alternating current brain stimulation (tACS) in neurodegenerative diseases. The investigators will evaluate whether a 4-times daily repeated stimulation with gamma tACS on the posterior parietal cortex can improve symptoms in patients with neurodegenerative diseases, including dementia with Lewy Bodies, Alzheimer's disease, idiopathic normal pressure hydrocephalus and Frontotemporal dementia.

ELIGIBILITY:
Inclusion Criteria:

* Mild Cognitive Impairment due to Alzheimer's disease
* Dementia with Lewy Bodies
* Frontotemporal dementia
* Idiopathic normal pressure hydrocephalus (iNPH)

Exclusion Criteria:

* History of seizures
* Pregnancy
* Metal implants in the head (except dental fillings)
* Electronic implants (i.e. pace-maker, implanted medical pump)
* Age <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-11-21 (Actual); Primary Completion 2032-07 (Estimated); Study Completion 2032-07 (Estimated)

PRIMARY OUTCOMES:
Changes in Rey Auditory Verbal Learning Test score | Baseline (immediately before the intervention), immediately after the first intervention, immediately after the 4th intervention, 4 weeks after the last intervention
  Participants are given a list of 15 unrelated words repeated over five different trials and are asked to repeat. Another list of 15 unrelated words are given and the patient must again repeat the original list of 15 words and then again after 30 minutes.
  The examiner reads aloud 15 unrelated words and the participant is asked to recall the words after each of the five trials. After a 15 minute delay, the participant is asked again to recall the words. The score ranges from 0 (worst performance) to 75 (best performance).
Changes in Rey Auditory Verbal Learning Test, recognition | Baseline (immediately before the intervention), immediately after the first intervention, immediately after the 4th intervention, 4 weeks after the last intervention
  Participants are given a list of 15 unrelated words repeated over five different trials and are asked to repeat.
  After a 15 minute delay, the participant is asked to recognise the original 15 words intermixed with 31 distractor words. The score of the recognition part ranges from 0 (worst performance) to 46 (best performance).
Changes in orientation to time and place (MMSE questions 1-10) | Baseline (immediately before the intervention), immediately after the last intervention, 4 weeks after the last intervention
  10 questions about the orientation. The score ranges from 0 (worse performance) to 10 (best performance).
Changes in Trail Making A & B tests | Baseline (immediately before the intervention), immediately after the 4th intervention, 4 weeks after the last intervention
  TMT A & B tests. Time to perform set is recorded.
Changes in INECO Frontal Screening test | Baseline (immediately before the intervention), immediately after the 4th intervention, 4 weeks after the last intervention
  Test battery assessing frontal lobe functions. The score ranges from 0 (worse performance) to 30 (best performance)
Changes in phonemic fluency | Baseline (immediately before the intervention), immediately after the first intervention, immediately after the 4th intervention, 4 weeks after the last intervention
  Person is requested to provide as many words as possible starting with certain letter. The score is the sum of all acceptable words produced in one minute.

SECONDARY OUTCOMES:
Change in SAI measurements | Baseline (immediately before the intervention), immediately after the last intervention
  By using transcranial magnetic stimulation (TMS), the investigators will evaluate the effects of gamma tACS on short latency afferent inhibition (SAI), which is a marker of cholinergic neurotransmission.
Change in SICI measurements | Baseline (immediately before the intervention), immediately after the last intervention
  By using transcranial magnetic stimulation (TMS), the investigators will evaluate the effects of gamma tACS on short interval intracortical inhibition (SICI), which is a marker of gabaergic neurotransmission.
Change in ICF measurements | Baseline (immediately before the intervention), immediately after the last intervention
  By using transcranial magnetic stimulation (TMS), the investigators will evaluate the effects of gamma tACS on intracortical facilitation (ICF), which is a marker of glutamatergic neurotransmission.

CONTACTS AND LOCATIONS:
Overall Officials: Eino Solje, MD, PhD, Principal Investigator — Kuopio University Hospital
Locations (1):
- Kuopio University Hospital, Kuopio, Finland

IPD SHARING:
Plan to Share IPD: Yes
Pseudonymized data upon request, according to Finnish national and EU GDPR regulations
Time Frame: Data will be shared after the study completion indefinitely.
Access Criteria: Reasonable request